CLINICAL TRIAL: NCT07235202
Title: An Open-label, Dose-escalation and Dose-expansion Phase Ib/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of MR001 in Combination With Standard Chemotherapy Regimens in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma (PDAC) Who Have Progressed After First-line Therapy
Brief Title: A Study of MR001 Combined With Chemotherapy in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma (PDAC) After First-line Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Majory Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MJR-MR001-02
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: MR001; PDAC; CD4; TGF-β1
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose Escalation Part1, Dose Group 1: MR001+Irinotecan Liposome+LV/5-FU (Experimental): MR001, 2mg/kg, QW; Irinotecan Liposome+LV/5-FU, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Irinotecan Liposome Injection combined with 5-FU/LV
- Dose Escalation Part1, Dose Group 2: MR001+Irinotecan Liposome+LV/5-FU (Experimental): MR001, 4mg/kg, QW; Irinotecan Liposome+LV/5-FU, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Irinotecan Liposome Injection combined with 5-FU/LV
- Dose Escalation Part1, Dose Group 3: MR001+Irinotecan Liposome+LV/5-FU (Experimental): MR001, 6mg/kg, QW; Irinotecan Liposome+LV/5-FU, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Irinotecan Liposome Injection combined with 5-FU/LV
- Dose Escalation Part2, Dose Group 1: MR001+nab-paclitaxel+gemcitabine (Experimental): MR001, 2mg/kg, QW; nab-paclitaxel+gemcitabine, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Nab-paclitaxel; Drug: Gemcitabine (GEM)
- Dose Escalation Part2, Dose Group 2: MR001+nab-paclitaxel+gemcitabine (Experimental): MR001, 4mg/kg, QW; nab-paclitaxel+gemcitabine, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Nab-paclitaxel; Drug: Gemcitabine (GEM)
- Dose Escalation Part2, Dose Group 3: MR001+nab-paclitaxel+gemcitabine (Experimental): MR001, 6mg/kg, QW; nab-paclitaxel+gemcitabine, Per locally approved dosage and administration
  Interventions: Drug: MR001; Drug: Nab-paclitaxel; Drug: Gemcitabine (GEM)
- Dose Expansion Part (Experimental): Based on the Dose escalation part results, the Investigator and Sponsor will determine one dose and dosing interval to proceed to the dose expansion study
  Interventions: Drug: MR001; Drug: Irinotecan Liposome Injection combined with 5-FU/LV; Drug: Nab-paclitaxel; Drug: Gemcitabine (GEM)

INTERVENTIONS:
Drug: MR001 — Intravenous infusion
Drug: Irinotecan Liposome Injection combined with 5-FU/LV — Per locally approved formulation
  Arms: Dose Escalation Part1, Dose Group 1: MR001+Irinotecan Liposome+LV/5-FU; Dose Escalation Part1, Dose Group 2: MR001+Irinotecan Liposome+LV/5-FU; Dose Escalation Part1, Dose Group 3: MR001+Irinotecan Liposome+LV/5-FU; Dose Expansion Part
Drug: Nab-paclitaxel — Per locally approved formulation
  Arms: Dose Escalation Part2, Dose Group 1: MR001+nab-paclitaxel+gemcitabine; Dose Escalation Part2, Dose Group 2: MR001+nab-paclitaxel+gemcitabine; Dose Escalation Part2, Dose Group 3: MR001+nab-paclitaxel+gemcitabine; Dose Expansion Part
Drug: Gemcitabine (GEM) — Per locally approved formulation
  Arms: Dose Escalation Part2, Dose Group 1: MR001+nab-paclitaxel+gemcitabine; Dose Escalation Part2, Dose Group 2: MR001+nab-paclitaxel+gemcitabine; Dose Escalation Part2, Dose Group 3: MR001+nab-paclitaxel+gemcitabine; Dose Expansion Part

SUMMARY:
This Phase Ib/IIa study is evaluating the safety, tolerability, pharmacokinetics, and preliminary efficacy of MR001 Combined with Chemotherapy in patients with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) who have progressed after first-line therapy.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation and dose-expansion Phase Ib/IIa study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of MR001 in combination with standard chemotherapy regimens in patients with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) who have progressed after first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic PDAC, progressed after only one prior line of systemic therapy.
* At least one measurable lesion per RECIST v1.1.
* ECOG Performance Status of 0-1.
* Life expectancy >3 months.
* Adequate organ and marrow function as defined by laboratory parameters.
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Known hypersensitivity to MR001 or similar monoclonal antibodies.
* Requirement for systemic immunosuppressive therapy within 14 days before first dosing.
* Uncontrolled active infections or concurrent malignancies.
* Not adequately controlled active brain metastases or leptomeningeal metastasis.
* Clinically significant cardiovascular, renal, or hepatic disorders.
* Pregnant or breastfeeding women.
* Any other circumstances which the investigator considers may increase risks to subjects or interfere with the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2028-06-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more dose-limiting toxicities (DLTs) | Approximately 12 months
Maximum Tolerated Dose (MTD) of MR001 | Approximately 12 months
  The maximum tolerated dose (MTD) of MR001 was assessed for QW dosing schedules
Incidence of Adverse Events (AEs) as Assessed by CTCAE v5.0 | Approximately 30 months
Objective Response Rate (ORR) | Approximately 24 months
Best Overall Response (BOR) | Approximately 24 months
Disease control rate (DCR) | Approximately 24 months

SECONDARY OUTCOMES:
Recommended Phase II Dose (RP2D) of MR001 in combination with standard chemotherapy regimens in patients with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) | Approximately 12 months
Progressionfree survival (PFS) | Approximately 24 months
Overall survival (OS) | Approximately 30 months
Area Under the Plasma ConcentrationTime Curve (AUC) of MR001 | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Maximum Plasma Concentration (Cmax) of MR001 | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Half-life (T1/2) of MR001 | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Incidence of Antidrug Antibodies (ADA) to MR001 | Predose in every 4 cycles for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Change from baseline at different time points for Th1 in plasma | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Change from baseline at different timepoints for Th2 in plasma | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Change from baseline at different timepoints for TGF-β1 in plasma | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)
Change from baseline at different time points for CD4 in plasma | Predose and at designated timepoints in each cycle for approximately 18 months (each cycle = 2 weeks or 4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No